CLINICAL TRIAL: NCT05916911
Title: Evaluación de la Eficacia de la combinación de GLIZIGEN® solución Oral 1/día y Gel Vaginal 1/Noche Durante 2 Meses en Pacientes Con Neoplasia Intraepitelial Cervical de Grado 1 (LSIL/CIN-1) Causada Por el Virus Del Papiloma Humano de Alto Riesgo (VPH-AR).
Brief Title: Evaluation Of The Efficacy Of The Combination Of GLIZIGEN® Oral Solution 1/Day And Vaginal Gel 1/Night For 2 Months In Patients With Cervical Intraepithelial Neoplasia Grade 1 (LSIL/CIN-1) Caused By High-Risk Human Papillomavirus (HPV-AR)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Collaborators: Atika Pharma S.L. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GLI-112
Record Dates: First submitted 2023-06-05; First posted 2023-06-23 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Papilloma Viral Infection; CIN1; LSIL, Low Grade Squamous Intraepithelial Lesion
Keywords: Glycyrrhizinic Acid; LSIL/CIN1; Cervical adenocarcinoma; Immunomodulation
MeSH Terms: conditions — Papillomavirus Infections; Squamous Intraepithelial Lesions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glizigen Group (Experimental): Patients will receive combined treatment with Glizigen® oral solution and Glizigen® vaginal gel for 2 months.
  Interventions: Dietary Supplement: Glizigen
- Placebo Group (Placebo Comparator): Patients will receive combined treatment with Placebo oral solution and Placebo vaginal gel for 2 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Glizigen — Treatment initiation: Treatment should be started simultaneously with the appropriate oral and intravaginal formulation after the last menstrual period or immediately in menopausal patients.
  A total of 60 single doses of intravaginal use and 60 doses of oral solution should be given to each patient.
  The intravaginal gel should be applied every night before going to sleep by inserting the cannula completely into the vagina and pressing the tube until the entire contents of the tube are poured into the vagina, then removing the cannula from the vagina while continuing to press the tube to avoid retrograde aspiration of the product. Application of the intravaginal gel should be discontinued during days of menstrual bleeding.
  The oral solution should be administered by drinking 1 vial every morning without interruption for 60 days from the start of treatment. It can be taken either on an empty stomach or with food.
  Arms: Glizigen Group
Other: Placebo — Treatment initiation: Treatment should be started simultaneously with the appropriate oral and intravaginal formulation after the last menstrual period or immediately in menopausal patients.
  A total of 60 placebo single doses of intravaginal use and 60 placebo doses of oral solution should be given to each patient.
  The placebo intravaginal gel should be applied every night before going to sleep by inserting the cannula completely into the vagina and pressing the tube until the entire contents of the tube are poured into the vagina, then removing the cannula from the vagina while continuing to press the tube to avoid retrograde aspiration of the product. Application of the intravaginal gel should be discontinued during days of menstrual bleeding.
  The placebo oral solution should be administered by drinking 1 vial every morning without interruption for 60 days from the start of treatment. It can be taken either on an empty stomach or with food.
  Arms: Placebo Group

SUMMARY:
HPV infection can lead to cancer, especially when precancerous lesions have developed and high-risk HPV is present.

Glizigen is an oral and intravaginal treatment based on activated glycyrrhizinic acid that has shown potential benefit in patients with HPV.

In order to improve the existing evidence, the present study consists of a randomized, double-blind, placebo-compared clinical trial to evaluate the efficacy of combined treatment with Glizigen Oral Solution and Glizigen Vaginal Gel for the resolution of biopsy-confirmed grade 1 cervical intraepithelial neoplasia (CIN-1) in patients with high-risk HPV.

DETAILED DESCRIPTION:
Human Papillomaviruses are double-stranded DNA viruses characterised by their lack of a lipid envelope. To date, more than 100 different types of HPV have been identified. They can be divided into cutaneous or mucosal depending on the tissues they usually infect 1. In parallel, HPVs can be classified as low-risk (HR-HPV) or high-risk (HR-HPV) viruses, depending on the risk of developing cancer due to their persistence of infection 2. Fifteen HPV types are considered high-risk (16, 18, 31, 33, 35, 35, 39, 45, 51, 52, 56, 58, 59, 68, 73 and 82) while three other types are classified as probable high-risk (26, 53 and 66).

HPV infection occurs through direct contact with the skin or mucous membranes of an infected person, who may or may not have visible lesions. In the case of genital infection, vaginal or anal intercourse is the main route of transmission. HPV is very common, and it is estimated that, in the United States, approximately 80% of women will have acquired an infection by the age of 50.

Most HPV infections do not cause symptoms or disease and disappear 12-24 months after infection. The small proportion of these infections that persist result in precancerous lesions that may progress to cancer. HPV infection is associated with virtually 100% of cervical cancer cases and with a high rate of anogenital and oropharyngeal cancers.

According to the World Health Organisation, the approach to cervical cancer prevention consists of primary prevention through HPV vaccination to prevent HPV infection, and secondary prevention through screening programmes to achieve early detection of HPV infection. Screening programmes differ from country to country, but are mainly based on determination of the presence of the virus by viral DNA testing and determination of intraepithelial lesions by cytology (Pap smear). A positive HPV DNA test implies the presence of the virus in the sample, while positive cytology implies an alteration or lesion in the tissue.

The morphology of squamous intraepithelial lesions caused by HPV in the lower anogenital tract is identical in all locations and in both sexes. The LAST Terminology classifies HPV-associated histological squamous intraepithelial lesions into two grades, low-grade lesions (LSIL) and high-grade lesions (HSIL). The term LSIL also includes cervical intraepithelial neoplasia grade 1 (CIN1) of the Richart classification, adopted by WHO in 2004.

LSIL/CIN1 lesions are the histological manifestation of a self-limiting HPV infection that most often resolves spontaneously. Close follow-up of patients with LSIL lesions minimises the risk of developing cervical cancer by observing whether the lesions resolve or, conversely, detecting early if they progress to HSIL. CIN2 and CIN3 lesions are included in the term HSIL. HSIL/CIN2 lesions can still revert to L-SIL or progress to neoplasia. In contrast, HSIL/CIN3 lesions are considered true intraepithelial neoplasms with a high potential for progression and are the necessary precursor lesion to cervical cancer and should be treated by destructive or excisional methods.

Another relatively common cytological alteration is atypical squamous cells of undetermined significance (ASCUS). An ASCUS cytology result may be due to HPV infection or other causes, so when detected, HPV-DNA testing is recommended. ASCUS is usually associated with SIL lesions, mainly LSIL, although HSIL cannot be ruled out.

On the other hand, colposcopy is an essential examination in the secondary prevention of cervical cancer (CCU) as it is the only procedure that allows the identification of intraepithelial cervical lesions, their location, extension and characteristics, and directs the biopsy to obtain diagnostic confirmation.

As previously advanced, secondary prevention is useful for early diagnosis of HPV infections, allowing treatment of high-grade lesions (HSIL) before they progress to cervical cancer. At the same time, it allows close follow-up of patients with low-grade lesions (LSIL). However, there is currently no specific treatment for LSILs, so it is limited to "wait and see" or observation without treatment.

Adequate nutritional status of patients with HPV infections is essential for optimal immune system function. Therefore, maintaining an adequate diet, smoking cessation and regular exercise are recommended as part of observational management strategies for patients with HPV infections. In some cases, supplementation of relevant macro- and micronutrients may help to stimulate the immune system and accelerate HPV clearance and lesion resolution. Indeed, dietary deficiencies of nutrients such as folates, vitamin C, vitamin B12, zinc and others have been linked to increased persistence of HPV infections and progression of HPV-related lesions. Moreover, other bio-functional ingredients with immunomodulatory, antiviral or antiproliferative activity could be useful both orally and topically.

Glizigen® vaginal gel and Glizigen® oral solution contain glycyrrhizinic acid as a common ingredient. Glycyrrhizinic acid or glycyrrhizin is a natural triterpenoid from liquorice root (Glycyrrhiza glabra) whose topical and systemic use has been evaluated in a multitude of studies that have demonstrated its safety and efficacy against different viral processeS. Among its most studied properties are its antiviral, anticarcinogenic and immunomodulatory action, and it has also been shown to have re-epithelialising, antibacterial, anti-inflammatory and antioxidant properties.

The mechanisms of antiviral action described for glycyrrhizinic acid against different viruses include: direct inactivation of the virus, reduction of virus fusion with the cell membrane, inhibition of viral replication, modulation of the immune response and stimulation of apoptosis:

In addition, glycyrrhizinic acid has demonstrated antiproliferative action against different types of cell lines or animal models of cervical, skin, colon or ovarian cancer. Specifically, it has been shown to be able to induce apoptosis and arrest the cell cycle in the G0/G1 phase in cervical cancer cells. Furthermore, it has a synergistic effect with cisplatin and 5-fluorouracil (5-FU) when combined with them. However, unlike cisplatin and 5-FU, glycyrrhizinic acid has no cytotoxic action against non-cancerous cells. Therefore, all these properties described for glycyrrhizinic acid make it a perfect candidate to prevent the proliferation of HPV-associated precancerous lesions.

Topical and systemic use of glycyrrhizinic acid activated by a catalytic process (Glizigen®) has been evaluated in women with HPV infections of the cervix, vagina or vulva, as well as in women and men with anogenital condylomas. The use of these formulations with activated glycyrrhizinic acid has shown good efficacy in favouring HPV negativisation and resolution of low-grade lesions (LSIL). It has also demonstrated a good safety profile and significantly superior efficacy to placebo and slightly superior efficacy to podophyllotoxin in the treatment of anogenital condylomata.

Rationale for the study HR-HPV infection carries a risk of developing cervical cancer, especially when precancerous lesions have already developed. The current screening system allows us to identify these patients; however, there is still no clear therapeutic option to treat patients before they develop high-grade lesions, where the most common management is surgical treatment.

Previous studies with Glizigen® provide evidence of its potential benefit in patients with cervical HPV infections, but there are a number of limitations that need to be addressed. Among them, the main limitation is that they are open-label, uncontrolled studies. It is true that Glizigen® has been used in comparative studies against placebo or podophyllotoxin in patients with anogenital condylomas . On the other hand, these studies in patients with HPV in the cervix included patients with both high- and low-risk HPV infection, who may or may not have histological lesions.

Therefore, this study would be justified by the following points:

* There is a need to investigate new therapeutic options, as there is no approved treatment for CIN1 lesions caused by HPV. It is therefore of interest to evaluate the efficacy of Glizigen® in the group of patients with HR-HPV LSIL/CIN1.
* It is of interest to evaluate the efficacy of the topical and systemic combination of Glizigen® with the new topical formulation.
* There is a need to provide higher quality evidence on the efficacy of Glizigen® than is currently available.

ELIGIBILITY:
Inclusion Criteria:

1. Women between 30 and 65 years of age.
2. Diagnosed with infection with at least one high-risk HPV strain (16, 18, 26, 31, 33, 35, 39, 45, 51, 52, 53, 56, 58, 59, 66, 68, 73 and 82) by PCR test and positive cytology with confirmation of LSIL/CIN-1 by colposcopy and biopsy.
3. Adequate cultural level and understanding of the clinical study.
4. Agree to participate voluntarily in the study and give written informed consent.

Exclusion Criteria:

1. Failure to meet any of the inclusion criteria.
2. Patient receiving any other product aimed at favouring the resolution of HPV infection.
3. Women with polymenorrhoea or frequent bleeding that makes vaginal administration of the preparation impossible.
4. Patient with immunosuppressive treatment or with other infectious processes in the genitals (e.g. herpes, candida, etc.).
5. Pregnant patients.
6. Participation in a concomitant trial that conflicts with this study.
7. Women with HIV infection.
8. Patients allergic to any component of the investigational product.

Patients who have been vaccinated against HPV before or after the start of the study are eligible to participate in the study, and this should be correctly reflected in the Data Collection Notebook.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-06-04 (Estimated); Study Completion 2025-01-08 (Estimated)

PRIMARY OUTCOMES:
Rate of resolution of cervical intraepithelial neoplasia grade 1 (CIN-1) caused by High Risk Human Papillomavirus (HR-HPV). | 6 months
  To assess whether nutritional supplementation with Glizigen® oral solution in combination with topical intravaginal use of Glizigen® vaginal gel promotes resolution of grade 1 cervical intraepithelial neoplasia (CIN-1) caused by High-Risk Human Papillomavirus (HR-HPV) compared to placebo after two months of treatment and 4 months after the end of treatment. It will be measured by biopsy.

SECONDARY OUTCOMES:
Antiviral effectiveness of glizigen against high-risk HPV infection. | 2 and 6 months
  To evaluate the efficacy of Glizigen® in improving the negativation rate of high-risk HPV strains (16, 18, 26, 31, 33, 35, 39, 45, 51, 52, 53, 56, 58, 59, 66, 68, 73 and 82) compared to placebo after two months of treatment and 4 months after the end of treatment by PCR.
Antiviral effectiveness of glizigen against multi high-risk HPV infection. | 2 and 6 months
  To assess the efficacy of Glizigen® in improving the negative rate of single or multiple high-risk HPV infections compared to placebo after two months of treatment and 4 months after the end of treatment by PCR.
Control of progression of Cervical intraepithelial neoplasia from CIN-1 to HSIL/CIN-2/3. | 2 and 6 months
  To evaluate the efficacy of Glizigen® in preventing the progression of cervical intraepithelial neoplasia from grade 1 (CIN-1) to grade 2 or 3 (HSIL/CIN-2/3) by colposcopy.
Grade of safety control | 2 and 6 months
  Assess safety at both systemic and local levels using treatment-related adverse effect monitoring questionnaires (YES/NO)
To Assess patient Tolerance of the study product. | 2 and 6 months
  To assess the patient's acceptance of the investigational product, questionnaires will be carried out during follow-up medical visits. Questionnaires are:
  - Tolerance questionnaire (YES/NO).
To Assess patient acceptance of the study product. | 2 and 6 months
  To assess the patient's acceptance of the investigational product, questionnaires will be carried out during follow-up medical visits. Questionnaires are:
  - Product acceptance questionnaire (YES/NO).
To Assess patient adherence of the study product. | 2 and 6 months
  To assess the patient's acceptance of the investigational product, questionnaires will be carried out during follow-up medical visits. Questionnaires are:
  - Treatment adherence questionnaire (YES/NO).
To Assess adherence to treatment | 2 and 6 months
  Assess adherence to treatment by following patients throughout the trial, calculating the average number of patients who stop treatment over the 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Pluvio J. Coronado Martín, Dr., Principal Investigator — Hospital San Carlos, Madrid
Locations (4):
- Spain (4):
  - Hospital Ruber Internacional, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Jung WW, Chun T, Sul D, Hwang KW, Kang HS, Lee DJ, Han IK. Strategies against human papillomavirus infection and cervical cancer. J Microbiol. 2004 Dec;42(4):255-66. PMID 15650698
- [Background] Rositch AF, Koshiol J, Hudgens MG, Razzaghi H, Backes DM, Pimenta JM, Franco EL, Poole C, Smith JS. Patterns of persistent genital human papillomavirus infection among women worldwide: a literature review and meta-analysis. Int J Cancer. 2013 Sep 15;133(6):1271-85. doi: 10.1002/ijc.27828. Epub 2012 Oct 11. PMID 22961444
- [Background] Munoz N, Bosch FX, de Sanjose S, Herrero R, Castellsague X, Shah KV, Snijders PJ, Meijer CJ; International Agency for Research on Cancer Multicenter Cervical Cancer Study Group. Epidemiologic classification of human papillomavirus types associated with cervical cancer. N Engl J Med. 2003 Feb 6;348(6):518-27. doi: 10.1056/NEJMoa021641. PMID 12571259
- [Background] Baseman JG, Koutsky LA. The epidemiology of human papillomavirus infections. J Clin Virol. 2005 Mar;32 Suppl 1:S16-24. doi: 10.1016/j.jcv.2004.12.008. PMID 15753008
- [Background] Braaten KP, Laufer MR. Human Papillomavirus (HPV), HPV-Related Disease, and the HPV Vaccine. Rev Obstet Gynecol. 2008 Winter;1(1):2-10. PMID 18701931
- [Background] de Sanjose S, Brotons M, Pavon MA. The natural history of human papillomavirus infection. Best Pract Res Clin Obstet Gynaecol. 2018 Feb;47:2-13. doi: 10.1016/j.bpobgyn.2017.08.015. Epub 2017 Sep 6. PMID 28964706
- [Background] Bosch FX, Broker TR, Forman D, Moscicki AB, Gillison ML, Doorbar J, Stern PL, Stanley M, Arbyn M, Poljak M, Cuzick J, Castle PE, Schiller JT, Markowitz LE, Fisher WA, Canfell K, Denny LA, Franco EL, Steben M, Kane MA, Schiffman M, Meijer CJ, Sankaranarayanan R, Castellsague X, Kim JJ, Brotons M, Alemany L, Albero G, Diaz M, de Sanjose S; authors of ICO Monograph Comprehensive Control of HPV Infections and Related Diseases Vaccine Volume 30, Supplement 5, 2012. Comprehensive control of human papillomavirus infections and related diseases. Vaccine. 2013 Dec 31;31 Suppl 7(Suppl 7):H1-31. doi: 10.1016/j.vaccine.2013.10.003. PMID 24332295
- [Background] Comprehensive Cervical Cancer Control: A Guide to Essential Practice. 2nd edition. Geneva: World Health Organization; 2014. Available from http://www.ncbi.nlm.nih.gov/books/NBK269619/ PMID 25642554
- [Background] Chan CK, Aimagambetova G, Ukybassova T, Kongrtay K, Azizan A. Human Papillomavirus Infection and Cervical Cancer: Epidemiology, Screening, and Vaccination-Review of Current Perspectives. J Oncol. 2019 Oct 10;2019:3257939. doi: 10.1155/2019/3257939. eCollection 2019. PMID 31687023
- [Background] Darragh TM, Colgan TJ, Cox JT, Heller DS, Henry MR, Luff RD, McCalmont T, Nayar R, Palefsky JM, Stoler MH, Wilkinson EJ, Zaino RJ, Wilbur DC; Members of LAST Project Work Groups. The Lower Anogenital Squamous Terminology Standardization Project for HPV-Associated Lesions: background and consensus recommendations from the College of American Pathologists and the American Society for Colposcopy and Cervical Pathology. Arch Pathol Lab Med. 2012 Oct;136(10):1266-97. doi: 10.5858/arpa.LGT200570. Epub 2012 Jun 28. PMID 22742517
- [Background] Kaufman RH. Dysplasia and carcinoma in situ of the cervix. Clin Obstet Gynecol. 1967 Dec;10(4):748-84. No abstract available. PMID 4172733